CLINICAL TRIAL: NCT05583162
Title: Healthy Sport Project: "Recovery, Body Acceptance and Health in Young Athletes"
Brief Title: Healthy Sport Project; Preventing Eating Disorders in Sport
Acronym: HSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold University College (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Therese Fostervold Mathisen, Associate Professor, Ostfold University College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 277766
Record Dates: First submitted 2022-10-08; First posted 2022-10-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Eating Disorders; Body Dissatisfaction; Disordered Eating; Adolescent - Emotional Problem; Athletic Injuries
Keywords: eating disorders; disordered eating; body dissatisfaction; figure idealisation; mental health; prevention; athlete; sport; adolescent; elite sport
MeSH Terms: conditions — Feeding and Eating Disorders; Athletic Injuries; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A cohort of athletes receive intervention in this pilot study, and changes from pre to post intervention are evaluated
Masking Description: Masking is not performed in a one-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All pupils attending a Elite Sport Jr High School receive intervention
  Interventions: Behavioral: Healthy Sport Project

INTERVENTIONS:
Behavioral: Healthy Sport Project — 2 interactive information lectures (given per class of 30 pupils), and 4 interactive workshops (given to sex-homogenous groups of 10 pupils). One per week, a total of 6 weeks with intervention.
  Other Names: Sports Body Project

SUMMARY:
The "Healthy Sport Project" is an adapted program from the Body Project by prof Eric Stice, aiming to reduce body dissatisfaction and symptoms of disordered eating and eating disorders in adolescent elite athletes. This trial aim to evaluate the effect of the program using a one-arm pilot study design in 14 years age old athletes at a Norwegian Elite Sport Junior High School.

DETAILED DESCRIPTION:
Eating disorders (EDs) are serious illnesses with highest incidence in adolescents. Moreover, athletes have a higher frequency of symptoms of disordered eating (DE) and EDs than non-athletes. There are many reasons to this health issue, but body appearance pressure, competing in body mass sensitive sports, and comments on body appearance are important explanations. Few programs have proved effective in preventing DE and EDs in the general population, or in athletes specifically, and none is permanent operative in sports in Norway. Body Project by prof Eric Stice have proved effective in preventing body dissatisfaction, figure idealization and new onset of EDs in female adolescents above 15 years of age, and with body dissatisfaction, from the general population. A few attempts to adapt this program to female athletes, argue for a comparative positive effect. Three important elements to further address, are: 1) programs need also to be tested in males; 2) programs need to be tested in adolescents of younger age before the typical onset of an ED; and 3) programs need to be possible to administer by non-professionals.

In this study the research group aim to adapt and test the effect of the Body Project, by the pilot study the "Healthy Sport Project", in elite junior athletes attending specialized junior sport high schools (age 14). The final goal for this project group is to create an effective preventive program for body dissatisfaction and DE/EDs in young athletes of both sexes and in mixed sports, and which may be administered by the schoolteachers.

ELIGIBILITY:
Inclusion Criteria:

* pupil at the recruited Sport Jr High School

Exclusion Criteria:

* no informed consent from parents
* not willing to participate
* a diagnosis of an eating disorder and being under (or waiting for) treatment

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Based on gender identity
Enrollment: 73 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of Eating Disorder, Eating Disorder Questionnaire Short-form | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  9 Questions on eating restriction, on worries for body weight and appearance. Rated by number of days the different content has been relevant. By Fairburn and Beglin, 2008
Change in Body Acceptance, Body Acceptance Scale, version 2 | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  10 Questions on body acceptance, rated by a 5 point Likert Scale (never - always). By Halliwell et al 2017.
Change in symptoms of internalization of body figure ideals, SATAQ-4 | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  10 Questions from subscales of SATAQ-4 (thinness idealisation and muscularity idealization), rated by 5 point Likert Scale. By Schaefer et al 2015
Experiences from participating in the project | After intervention (post, +6 weeks)
  Focus group interview following a semistructured manual; asking for experiences with participation in the "Healthy Sport Project"

SECONDARY OUTCOMES:
Change in experiences of Body Appearance Pressure (BAP), questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Question on experience of BAP (if it is experienced yes/no)
Change in experiences of Body Appearance Pressure (BAP), questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Question on arenas for experience of BAP (in which contexts; choose between listed arenas)
Change in dietary habits, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Questions on meal frequency (numbers); frequency of intake of fruit and vegetables (number of portions); frequency of intake of dairy products (number of portions); frequency of intake of fish (number of portions)
Change in dietary habits, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Use of supplements (yes/no)
Change in dietary habits, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Use of supplements ( what type of supplements, chose from listed alternatives)
Change in nutrition knowledge, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  3 questions asking for examples of foods providing carbohydrates; proteins; fats, respectively.

OTHER OUTCOMES:
Question on injuries, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  1 Questions asking for any incident of injury (yes/no)
Question on injuries, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Where the injury was located (chose from list of anatomical locations)
Demographics, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Age (years)
Demographics, questions by research group | Before intervention
  Sex (male/female)
Demographics, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Sport (any given)
Demographics, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Body weight (kg)
Demographics, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Height (m)
Demographics, questions by research group | Before intervention, After intervention (post, +6 weeks), 6 months after end of intervention
  Number of hours in physical activity per week (hours).

CONTACTS AND LOCATIONS:
Overall Officials: Therese F Mathisen, PhD, Principal Investigator — Østfold University College
Locations (1):
- Therese Fostervold Mathisen, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No
Not to be shared